CLINICAL TRIAL: NCT06761417
Title: A Prospective, Single-arm Clinical Study of Liposomal Mitoxantrone Combination Regimen in the Treatment of Relapsed and Refractory Solid Tumors in Children, Adolescents and Young Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, SIDAN LI, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5006
Record Dates: First submitted 2024-12-29; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors; Children; Adolescents
Keywords: Mitoxantrone liposomes; Solid tumor; Children and adolescents
MeSH Terms: interventions — Capecitabine; anlotinib

STUDY DESIGN:
Intervention Model Description: It is expected to enroll 49 patients with relapsed and refractory solid tumors in children, adolescents and young adults. The treatment will be carried out using the liposomal mitoxantrone combination regimen. The minimum acceptable objective response rate (ORR) is 30%, and the expected ORR is 50%. The study includes a screening period (within 28 days), a treatment period (planned for 6 cycles), and a follow-up period (safety follow-up and progression-free survival (PFS) follow-up). Subjects who sign the informed consent form and undergo baseline examinations within the screening period, and those who meet the inclusion and exclusion criteria will enter the treatment period, with one cycle every 3 weeks. All subjects will complete the relevant examinations specified in the protocol during the treatment process to observe the safety and efficacy. After the treatment period, they will enter the follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal Mitoxantrone Combination Regimen (Experimental): Mitoxantrone liposome+Capecitabine+Anlotinib
  Interventions: Drug: Mitoxantrone liposome; Drug: Capecitabine; Drug: Anlotinib

INTERVENTIONS:
Drug: Mitoxantrone liposome — Mitoxantrone liposome: 16 mg/m^2, d1; Each 21-day cycle was used for a total of 4-6 cycles.
Drug: Capecitabine — Capecitabine 1000 mg/m^2, d1-14, bid; Each 21-day cycle was used for a total of 4-6 cycles.
Drug: Anlotinib — Anlotinib: according to patient weight: 8mg/ day in patients <35kg; 10mg/ day for patients with 35kg≤ patient weight ≤50kg; 12mg/ day for patients > 50kg; d1-14; Each 21-day cycle was used for a total of 4-6 cycles.

SUMMARY:
The aim of this clinical study is to determine the efficacy and safety of the liposomal mitoxantrone combination regimen in treating relapsed and refractory solid tumors among children, adolescents, and young adults. The key questions it intends to address are:

Can the liposomal mitoxantrone combination regimen improve the objective response rate (ORR) compared to historical data? What are the adverse events associated with this combination regimen? Researchers will administer the liposomal mitoxantrone combination regimen (including capecitabine and anlotinib with specific dosing regimens) to the participants and closely monitor their conditions.

Participants will:

Receive the treatment regimen for 4 - 6 cycles, with each cycle lasting 21 days Undergo regular checkups and tests during the treatment period and follow-up period as per the protocol.

Have their tumor status, blood parameters, and other relevant indicators measured to evaluate the treatment effect and safety.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter clinical study named "A Prospective, Single-arm, Multicenter Clinical Study of Liposomal Mitoxantrone Combination Regimen in the Treatment of Relapsed and Refractory Solid Tumors in Children, Adolescents and Young Adults". The study aims to assess the safety and effectiveness of the liposomal mitoxantrone combination regimen in treating relapsed and refractory solid tumors among children, adolescents, and young adults.

The research anticipates enrolling 49 patients meeting specific criteria. The inclusion criteria require patients to have a clear understanding of the study, sign the informed consent form voluntarily, fall within the age range of 6 - 24 years with an expected survival time exceeding 3 months, have histopathologically confirmed relapsed and refractory solid tumors of certain subtypes (such as bone and soft tissue tumors, neuroblastoma, etc.), possess measurable tumor lesions detectable by CT, enhanced CT, PET/CT or MRI, and meet specific Karnofsky and ECOG scores as well as requirements for bone marrow, liver, and kidney functions. Exclusion criteria cover those with hypersensitivity to study drugs, uncontrolled other malignancies, pregnant or lactating women, and those judged unsuitable by investigators.

The treatment regimen consists of capecitabine at a dose of 1000 mg/m² from day 1 to 14, twice daily, and anlotinib with the dose adjusted according to body weight for 14 days, with a 21-day cycle repeated 4 - 6 times. Patients achieving a partial response or better will undergo local treatment like surgery or radiotherapy.

The primary endpoint of the study is the objective response rate (ORR), while secondary endpoints include the proportion of patients eligible for local treatment after treatment, disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and adverse events evaluated by NCI CTCAE v5.0. This study holds great significance for exploring new treatment options for relapsed and refractory solid tumors in the target population.

ELIGIBILITY:
Main inclusion Criteria:

1. The patient fully understands this study, voluntarily participates and signs the informed consent form (ICF).
2. Age: children (6 - 12 years old), adolescents (13 - 18 years old) and young adults (19 - 24 years old) (CAYA). The expected survival time is > 3 months.
3. Diagnosed with relapsed and refractory solid tumors by histopathology, and it is one of the following subtypes: (1) bone and soft tissue tumors; (2) neuroblastoma; (3) other types of solid tumors that the investigator deems eligible for enrollment.
4. There must be measurable tumor lesions by CT, enhanced CT, PET/CT or MRI.
5. Karnofsky score > 50; ECOG score ≤ 2.
6. Bone marrow function: neutrophil count > 1.5 × 10⁹/L, platelet count > 75 × 10⁹/L, hemoglobin ≥ 80 g/L.
7. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and ALT < 2.5 times the upper limit of normal value (for patients with liver invasion < 5 times the upper limit of normal value); total bilirubin < 1.5 times the upper limit of normal value (for patients with liver invasion < 3 times the upper limit of normal value).
8. No history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, no history of clinically severe pericardial disease, or no electrocardiogram evidence of acute ischemic or active conduction system abnormality within 6 months before recruitment.

Main exclusion Criteria:

1. Patients with known hypersensitivity to any component of the study drugs.
2. Patients with other malignant tumors that are not under control (except for basal cell carcinoma of the skin, in-situ breast/cervical cancer, and other malignant tumors that have been effectively controlled without treatment in the past five years).
3. Pregnant, lactating women and women of childbearing age who are unwilling to take contraceptive measures.
4. Other situations judged by the investigator as not suitable for participating in this study.

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Objective response(ORR) | Up to 6 cycles of chemotherapy (each cycle is 21 days)
  Rate of Objective response (ORR) after 4 or 6 cycles of Liposomal Mitoxantrone Combination Regimen, including complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Rate of Disease control (DCR) | Up to 6 cycles of Liposomal Mitoxantrone Combination Regimen (each cycle is 21 days)
  Refers to the percentage of patients with confirmed complete response, partial response, and disease stability in patients with evaluable efficacy
Progression-free survival (PFS) | From date of enrollment unit the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  Means from the date of enrollment to the date of first disease progression or death from any cause, whichever comes first. If the subject has no disease progression during the trial period, PFS is defined as the last date until the subject's last confirmed progression-free survival.
Overall survival (OS) | From date of enrollment unit the date of first documented date of death from any cause, assessed up to 24 months.
  Overall survival (OS) was defined from the date of enrollment to the date of death from any cause.
Proportion of patients eligible for local treatment after treatment | Up to 6 cycles of chemotherapy (each cycle is 21 days)
  Proportion of patients who meet the conditions for local treatment after treatment. mathematically, it can be expressed as: Proportion = (Number of patients eligible for local treatment / Total number of patients in the study) × 100%.
Safty | After signing the informed consent form, the safety monitoring began and continued until the end of the follow-up (follow-up period of 1 year).
  Number of subjects with each adverse event. Safety Evaluation Criteria: The National Cancer Institute Adverse Event Common Terminology Criteria (NCICTCAE V.5.0) were used to judge the adverse events and severity during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No